CLINICAL TRIAL: NCT01276392
Title: Platelet Function, Whole Blood Coagulation and Fibrinolysis During Continuous Renal Replacement Therapy - a Comparison of Citrate and Heparin Anticoagulation
Brief Title: Anticoagulation and Activation - Comparison in Continuous Renal Replacement Therapy
Status: Withdrawn | Type: Observational
Why Stopped: A main person involved left the site
Sponsor: Klinik für Anästhesiologie (Other)
Responsible Party: Sponsor-Investigator, Klinik für Anästhesiologie, Leiter Interdisziplinäre Operative Intensivstation ZOM-I, Heinrich-Heine University, Duesseldorf
Organization: Heinrich-Heine University, Duesseldorf (Other)
Other Study IDs: 01-AHTSDKM
Record Dates: First submitted 2011-01-12; First posted 2011-01-13 (Estimated); Last update posted 2015-08-20 (Estimated); Status verified 2015-08

CONDITIONS: Kidney Replacement Disorder
Keywords: regional and systemical anticoagulation; continuous renal replacement therapy; multiplate; rotational thrombelastometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Heparin: 10 Patients undergoing continuous renal replacement therapy using heparin for providing anticoagulation. Blood samples taken at 8 predefined timepoints.
- CiCa: 10 Patients undergoing continuous renal replacement therapy using citrate for providing anticoagulation. Blood samples taken at 8 predefined timepoints.

SUMMARY:
Actual clinical practice predominantly makes use of heparin (systemically) or citrate regionally as anticoagulation in the extracorporeal circulation for renal replacement therapy. We aim to find out if different anticoagulation strategies may lead to different levels of platelet activation and whole blood coagulation. Regarding coagulation activation, it remains uncertain if there is an advantage for one of these methods. However, it is of major interest to minimize the risk of any additional clotting activation via extracorporeal circulation in these usually critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years, acute renal failure with need for continuous veno-venous renal replacement therapy

Exclusion Criteria:

* Age < 18 years, pregnancy, contraindications for one of the two anticoagulation methods, missing informed consent or disagreement in the progress of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critical ill patients with acute renal failure and the need of continuous renal replacement therapy.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2011-01; Primary Completion 2014-11 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
Filter life time of continuous renal replacement therapy | Individual time point, standardized
  Filter life time measured in hours of duration of continuos renal replacement therapy, filter life time end, when system clotts.

SECONDARY OUTCOMES:
Activation of coagulation | beginning of hemodialysis, 1,2,4,12,24,28,72 hours after start of hemodialysis
  blood samples for multiplate, rotem and systemic coagulation paramters

CONTACTS AND LOCATIONS:
Overall Officials: Detlev Kindgen-Milles, Professor,MD, Principal Investigator — Department of Anesthesiology, University Hospital Duesseldorf, Heinrich Heine University
Locations (1):
- Interdisciplinary Operative Intensive Care Unit, University Hospital Duesseldorf, Düsseldorf, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Schaefer RM, Barenbrock M, Teschner M, Bahner U. [Extracorporeal renal replacement therapies in acute renal failure]. Med Klin (Munich). 2000 May 15;95(5):273-8. doi: 10.1007/pl00002121. German. PMID 10850066
- [Background] Toft P, Gilsaa T. [Acute renal failure in critically ill patients]. Ugeskr Laeger. 2007 Feb 19;169(8):692-5. Danish. PMID 17313917
- [Background] Davenport A. The coagulation system in the critically ill patient with acute renal failure and the effect of an extracorporeal circuit. Am J Kidney Dis. 1997 Nov;30(5 Suppl 4):S20-7. doi: 10.1016/s0272-6386(97)90538-2. PMID 9372975
- [Background] Bouman CS, de Pont AC, Meijers JC, Bakhtiari K, Roem D, Zeerleder S, Wolbink G, Korevaar JC, Levi M, de Jonge E. The effects of continuous venovenous hemofiltration on coagulation activation. Crit Care. 2006;10(5):R150. doi: 10.1186/cc5080. PMID 17069648
- [Background] Sabovic M, Salobir B, Preloznik Zupan I, Bratina P, Bojec V, Buturovic Ponikvar J. The influence of the haemodialysis procedure on platelets, coagulation and fibrinolysis. Pathophysiol Haemost Thromb. 2005;34(6):274-8. doi: 10.1159/000093107. PMID 16772739
- [Background] Lang T, von Depka M. [Possibilities and limitations of thrombelastometry/-graphy]. Hamostaseologie. 2006 Aug;26(3 Suppl 1):S20-9. German. PMID 16953288